CLINICAL TRIAL: NCT03834233
Title: A Phase II of Study of Nivolumab in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Nivolumab in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Acronym: CA209-9JC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo R Munhoz, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1258/18
Record Dates: First submitted 2019-02-03; First posted 2019-02-07 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 3mg/kg IV every 14 days until disease progression, unacceptable toxicity or up to 12 months.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3mg/kg IV every 14 days until disease progression, unacceptable toxicity or up to 12 months.

SUMMARY:
Cutaneous squamous cell carcinoma (cSCC) is one of the most frequent malignancies worldwide, and an increasing incidence has been documented over the past decades. Despite optimal initial approach, which can be curative in the majority of cases, a proportion of patients present with locally advanced or unresectable disease, leading to significant morbidity. In addition, metastases of cSCC may affect 2 to 5% of individuals diagnosed with this disease. In the setting of advanced cSCC, no standard systemic treatment has been established, and treatment options are frequently adapted from those applied to squamous cell carcinoma arising from other sites, based on a low level of evidence and often with short-lived benefits.

cSCC are potentially immunogenic neoplasms with an unmet need for therapeutic options, having sun exposure and chronic inflammation as the most significant risk factors. Using the anti-PD1 monoclonal antibody nivolumab to treat patients with cSCC and planned scientific correlates, investigators believe that the safety and efficacy of immune activating therapy for this disease can be assessed.

This is a multi-center, Simon two-stage, phase II study to evaluate the safety and efficacy of the anti-PD1 monoclonal antibody nivolumab for systemic-treatment-naïve patients with metastatic and/or locally advanced cSCC.

The primary objective of the study is to evaluate the efficacy, as assessed by the best objective response rate (complete response + partial response) at 24 weeks according to RECIST criteria, of nivolumab in patients with advanced cSCC. Secondary objectives are to assess the safety/tolerability of the treatment, to determine the progression-free survival (PFS) and overall survival (OS) rates at 24 weeks, and to evaluate the objective response rate as assessed by immune-related response criteria (irRC). Treatment will be given every 14 days until disease progression, unacceptable toxicity or withdrawal of consent/patient decision. If the patient continues to benefit from treatment with nivolumab, treatment will be continued for up to 12 months. Patients will be reassessed at week 12 and every 12 weeks thereafter until week 52, and then as per discretion of the treating investigator. A tumor biopsy will be performed before treatment initiation, unless contraindicated and optional biopsies will be performed at week 13 and following disease progression. Serial blood samples will be obtained at baseline, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age.
* Subjects must have a histologically confirmed metastatic/locally advanced cutaneous squamous cell carcinoma
* No prior systemic treatments for advanced (metastatic or locally advanced) cSCC
* Measurable disease as defined by RECIST 1.1
* Performance status: ECOG 0 to 1
* Patients must be recovered from surgery or toxic effects of prior radiation therapy. Study treatment may not start until at least two weeks from completion of radiation therapy or surgery.
* Adequate hematologic, hepatic and renal function as defined below i. Hemoglobin > 8.5 g/dl (can be post transfusion) ii. Absolute neutrophil count > 1,000/mm3 iii. Platelet count > 75,000/mm3 iv. Total Bilirubin <2.0 x upper limit of normal (ULN) in absence of Gilbert disease (Total Bilirubin ≤ 3 x ULN with Gilbert).

  v. ALT (SGOT) or AST (SGPT) <2.0 x ULN (or < 3 times the upper limit of normal are permitted if clearly attributed to liver metastasis) vi. Calculated creatinine clearance (CrCI) ≥ 30 mL/min using the lean body mass formula only (Modified Cockroft and Gault; Shargel and Yu 1985)
* Ability to understand informed consent and comply with treatment protocol
* Male and female patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device [IUD], birth control pills, or barrier device) during and for 5 months (females) or 7 months (males) after the study. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 30 days prior to study enrollment. Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study and for 7 months following the last dose of study drug

Exclusion Criteria:

* Prior use of anti-PD-1 or anti-PD-L1 monoclonal antibody.
* Uncontrolled intercurrent illness including active infection or symptomatic congestive heart failure within 6 months
* Patients requiring systemic treatment with corticosteroids (>10mg daily of prednisone or equivalent) or using immunosuppressive medications within 10 days of study drug administration.
* Patients with untreated or symptomatic brain metastases.
* Known history of immunodeficiency virus disease with detectable viral load and CD4+ lymphocyte count <350 mm3. Patients with undetectable vital load and CD4+ lymphocyte count >350 mm3 are eligible
* History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or documented history of autoimmune disease or syndrome requiring systemic steroids or immunosuppressive agents except vitiligo or resolved childhood asthma/atopy.
* Evidence of clinically significant immunosuppression, including primary immunodeficiency state such as Severe Combined Immunodeficiency Disease or concurrent opportunistic infection
* Known active hepatitis B or hepatitis C infection. Patients with undetectable viral load for hepatitis B or C as determined by PCR are eligible.
* History of stem-cell or solid organ transplant.
* Received live vaccine within 28 days prior to enrollment
* Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 5 months after the last dose of nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate (complete response + partial response) using RECIST criteria at 24 weeks | From date of treatment initiation until week 24
  To evaluate the efficacy, as assessed by the best objective response rate (complete response + partial response) at 24 weeks by RECIST 1.1, of nivolumab in patients with advanced cSCC.

SECONDARY OUTCOMES:
Incidence of treatment related adverse events | From date of treatment initiation until week 24
  To assess the safety and tolerability of nivolumab in patients with advanced cSCC.
Progression free survival (PFS) rate | From date of treatment initiation until week 24
  To determine the progression free survival (PFS) rate at 24 weeks
Best objective response rate (complete response + partial response) using immune-related response criteria | From date of treatment initiation until week 24
  To evaluate the efficacy, as assessed by the best objective response rate (complete response + partial response) at 24 weeks by immune-related response criteria (irRC), of nivolumab in patients with advanced cSCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Ramella Munhoz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munhoz RR, Nader-Marta G, de Camargo VP, Queiroz MM, Cury-Martins J, Ricci H, de Mattos MR, de Menezes TAF, Machado GUC, Bertolli E, Barros M, de Souza CE, Franke F, Ferreira FO, Feher O, de Castro G Jr. A phase 2 study of first-line nivolumab in patients with locally advanced or metastatic cutaneous squamous-cell carcinoma. Cancer. 2022 Dec 15;128(24):4223-4231. doi: 10.1002/cncr.34463. Epub 2022 Oct 24. PMID 36274573